CLINICAL TRIAL: NCT06736067
Title: Effects of a Single-bout of Moderate-intensity Aerobic Exercise on Mood and Mental Health Biomarkers in Adults with Depressive And/or Anxiety Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YAU Suk Yu Sonata (Other)
Responsible Party: Sponsor-Investigator, YAU Suk Yu Sonata, Associate Professor, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSEARS20221111001-01
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Depression Symptoms; Anxiety Symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Moderate-intensity aerobic exercise (Experimental): Thirty minutes of exercise on a treadmill, including a 5-minute warm-up followed by increments in speed until reaching optimal moderate to high intensity (60-80% of age-predicted maximal heart rate), which will be maintained for 20 min, followed by a 5-minute cool-down. Age-predicted maximal HR will be defined as 220 beats-per-minute (BPM) minus age in years.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Thirty minutes of exercise on a treadmill, including a 5-minute warm-up followed by increments in speed until reaching optimal moderate to high intensity (60-80% of age-predicted maximal heart rate), which will be maintained for 20 min, followed by a 5-minute cool-down. Age-predicted maximal HR will be defined as 220 beats-per-minute (BPM) minus age in years.

SUMMARY:
This study investigates whether a single session of aerobic exercise (like running) can improve the participants' mood and whether such benefits can be explained by changes in the blood factors (like hormones) and brain activity.

The main questions this study aims to answer are:

* Can a single session of aerobic exercise improve mood?
* Which changes in the blood and brain could explain the effects of exercise on mood?

Researchers will compare the participants' mood states before and after exercise to see whether exercise can improve mood.

The participants will:

* Answer questionnaires, collect blood, and undergo magnetic resonance imaging (MRI) before exercise.
* Perform 30 minutes of running on a treadmill.
* Answer the same questionnaires, collect blood, and undergo magnetic resonance imaging (MRI) after exercise.

The entire assessment will last for about 2h45min and will be performed on a single day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects within the stipulated age range

Exclusion Criteria:

* Acute injury or illness that impairs the ability to safely exercise and/or inability to exercise with a moderate intensity;
* Metabolic and/or neurologic disorders;
* Iron implants;
* People who cannot stay still, are intolerant of noise or fearful of enclosed spaces (due to the small space inside the scanner).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | From before to immediately after a single session of exercise
  POMS is a 30-item questionnaire scored on a 5-point Likert-type scale ranging from "Not at all" to "Extremely." It provides six sub≥scales: 1) anger (e.g., grouchy, furious); 2) confusion (e.g., muddled, forgetful); 3) depression (e.g., sad, unworthy); 4) fatigue (e.g., tired, sluggish); 5) tension (e.g., nervous, anxious); and 6) vigor (e.g., lively, active).

SECONDARY OUTCOMES:
Subjective Exercise Experience Scale (SEES) | From before to immediately after a single session of exercise
  SEES is a 12-item questionnaire that is scored on a 7-point Likert-type scale ranging from "Not at all" to "Very much". It Provides 3 subscales that will be used in the present study: 1) psychological well-being (great, positive, strong, terrific); 2) psychological distress (awful, crummy, discouraged, miserable); and 3) fatigue (drained, exhausted, fatigued, tired).
Subject Happiness Scale (SHS) | From before to immediately after a single session of exercise
  SHS is a 4-item self-report measure developed to assess an individual's overall happiness as measured through self-evaluation. The response format is a 7-point Likert-type scale.
Blood biomarkers | From before to immediately after a single session of exercise
  Blood biomarkers, including brain-derived neurotrophic factor (BDNF) and Adiponectin
Cardiovascular parameters | Before, during, and immediately after a single session of exercise
  Heart Rate Variability (HRV) will be monitored during all the exercise protocol.
BOLD-weighted fMRI images | From before to immediately after a single session of exercise
  BOLD-weighted fMRI images will be acquired using a gradient-echo echo-planar imaging (GRE-EPI) sequence with (a) repetition time = 2000 ms, (b) echo time = 30 ms, (c) flip angle = 90°, (d) matrix = 64 × 64, (e) field of view = 220 mm × 220 mm, (f) slice thickness = 4 mm with interslice gap = 0.6 mm, and (g) 33 interleaved axial slices. Additionally, weighted images will be acquired with an interleaved sequence (188 sagittal slices, TR/TE/flip angle = 8.2 ms/3.7 ms/7°, matrix = 256 × 256 mm2, FOV = 256 × 256 × 188 mm, and voxel size = 1 × 1 × 1 mm3).
Diffusion-weighted image (DWI) | From before to immediately after a single session of exercise
  Whole-brain diffusion-weighted image (DWI) will be collected with a single-shot diffusion-weighted echo planar imaging sequence (TE, 83 ms; TR, 8700 ms; flip angle, 90°; image resolution, 1.64 mm isotropic; b value, 800 s/mm2; 70 axial slices) in 30 diffusion encoding directions and one non-diffusion-weighted reference image (b = 0).
Magnetic resonance spectroscopy (MRS) | From before to immediately after a single session of exercise
  Magnetic resonance spectroscopy (MRS) will be utilized to measure levels of glutamate and GABA.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided